CLINICAL TRIAL: NCT05892198
Title: A Single Center Experience in the Management of Pilonidal Disease; the Impact of Pits Location on the Choice of the Best Surgical Option.
Brief Title: A Single Center Experience in the Management of Pilonidal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmad Sakr, Lecturer of general surgery, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1122
Record Dates: First submitted 2023-05-28; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Pilonidal Sinus
Keywords: sacrococcygeal pilonidal sinus; primary closure; limberg flap; rotational flap
MeSH Terms: conditions — Pilonidal Sinus | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- primary closure (Active Comparator): The group in which the pits location were in midline ,underwent excision with primary closure
  Interventions: Procedure: surgery
- Rhomboid flap group (Active Comparator): in which more lateral pits and pits located <2cm from mid line natal cleft
  Interventions: Procedure: surgery
- Rotational flap group (Active Comparator): in which more lateral pits and pits located >2cm from mid line natal cleft
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — surgery with primary closure, Rhomboid flap , or Rotational flap
  Other Names: surgical procedure

SUMMARY:
Sacrococcygeal pilonidal disease (PND) is a common entity affecting the skin and subcutaneous tissue of the upper portion of the natal cleft of the buttocks. It is characterized by the presence of sinus tracts with recurrent inflammation and infection. It poses a significant healthcare problem due to its related morbidity, impaired quality of life, and financial costs.

DETAILED DESCRIPTION:
This acquired disease is caused by negative suction of the hair present in the natal cleft region, leading to a foreign body reaction and subsequent granuloma . It affects 26 per 100000 people, and it mainly affects young men . Surgery for PND is frequently performed in Egypt by general surgeons, with no published data regarding its incidence or prevalence in the Egyptian population.

The PND patient may report different presentations ranging from asymptomatic disease to acute infection and abscess formation. Others may have a chronic disease with recurrent perianal inflammation and discharge.

Multiple surgical options have been described for chronic PND. However, no technique has been universally accepted. The idea of any procedure is to excise the pits with the related sinus tracts leaving healthy tissue as possible to decrease recurrence. The most commonly performed surgical techniques include excision with either primary closure, lay open, or flap-based reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes
* aging between 18- 60 years old
* who underwent surgical intervention for the pilonidal sinus (Either primary or recurrent)
* The surgical intervention includes excision with primary closure or lay open technique, Rhomboid flap and rotational flap.

Exclusion Criteria:

* surgically unfit due to commodities.
* those who lost follow up

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Select the best operative technique as regard the number and distribution of the pits in pilonidal sinus cases. | 6 months
  best surgical option based on pits location
Recurrence rate | 6 months - 1 year
  how many cases developed recurrence

SECONDARY OUTCOMES:
the incidence of complications such as: wound infection, wound dehiscence, postoperative pain. | 1 month
  complication rate

IPD SHARING:
Plan to Share IPD: No